CLINICAL TRIAL: NCT00884819
Title: Effects of Fenofibrate on Metabolic and Reproductive Parameters in Polycystic Ovary Syndrome. A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of Fenofibrate on Metabolic and Reproductive Parameters in Polycystic Ovary Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tisha Joy, Assistant Professor, Division of Endocrinology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-08-573; 15581 (Other: UWO Ethics)
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; hepatic adiposity; diabetes; hormones; cardiovascular disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Diabetes Mellitus; Cardiovascular Diseases | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): fenofibrate 200mg/daily for 6 months
  Interventions: Drug: Fenofibrate
- 2 (Placebo Comparator): Placebo match for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fenofibrate — fenofibrate 200 mg daily for 6-months
  Arms: 1
Other: Placebo — Placebo match for 6 months
  Arms: 2

SUMMARY:
This is a prospective randomized, double-blind placebo-controlled trial of 6 months' duration evaluating the effect of fenofibrate (200 mg/day) in females with polycystic ovary syndrome and mild hypertriglyceridemia. The investigators primary objective will be to determine whether fenofibrate will reduce hepatic adiposity as measured using MRI, and our secondary outcomes will be to delineate the impact of fenofibrate on biochemical or clinical parameters for insulin resistance, cardiovascular disease, and reproductive status.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal women ≥ 18 years
* diagnosis of PCOS based on the recent 2006 Androgen Excess Society criteria (modified from Rotterdam 2003)
* waist circumference >88 cm
* fasting TG 2.0 - 5.0 mmol/L
* stable on any type of oral contraceptive for a minimum of 3-months

Exclusion Criteria:

* known contraindications for MRI
* pregnancy, lactation, desire to become pregnant
* participation in another clinical trial
* fasting TF level ≥ 5.0 mmol/L
* AST or ALT > 2.5 times upper limit of normal (ULN)
* creatinine kinase (CK) > 6x ULN
* creatinine > 115 μmol/L
* fasting glucose ≥ 7.0 mmol/L and/or 2h glucose post oral glucose tolerance test (OGTT) ≥ 11.1 mmol/L or personal history of DM2
* personal history of renal disease, liver disease (except NAFLD), or heart disease
* body mass index (BMI) < 18 or > 40 kg/m²
* increased alcohol use (>9 standard drinks per week [standard drink = 12oz beer, 5oz wine, or 1.5oz spirits]) or drug use
* use of other hormonal contraception, growth hormone, glucocorticoids, anti-diabetic/anti-dyslipidemia medications, or anabolic steroids.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Hepatic adiposity as assessed using MRI | 6-months

SECONDARY OUTCOMES:
Body composition using bioelectrical impedance analysis (BIA), anthropometry (skin-fold thickness measurement), and MRI | 6-months
Insulin resistance using HOMA-IR | 6 months
Biochemical parameters related to insulin resistance (adipocytokines, free fatty acids, 25-hydroxyvitamin D) | 6 months
Traditional and non-traditional cardiovascular risk factors (lipids, apolipoproteins, fibrinogen, PAI-1, CRP) | 6 months
Reproductive parameters (androgens, hirsutism) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tisha Joy, MD FRCPC, Principal Investigator — St. Joseph's Health Care, Department of Medicine
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Toda K, Okada T, Miyaura C, Saibara T. Fenofibrate, a ligand for PPARalpha, inhibits aromatase cytochrome P450 expression in the ovary of mouse. J Lipid Res. 2003 Feb;44(2):265-70. doi: 10.1194/jlr.M200327-JLR200. Epub 2002 Nov 4. PMID 12576508
- [Background] Wysocki J, Belowski D, Kalina M, Kochanski L, Okopien B, Kalina Z. Effects of micronized fenofibrate on insulin resistance in patients with metabolic syndrome. Int J Clin Pharmacol Ther. 2004 Apr;42(4):212-7. doi: 10.5414/cpp42212. PMID 15124979
- [Background] Lee HJ, Choi SS, Park MK, An YJ, Seo SY, Kim MC, Hong SH, Hwang TH, Kang DY, Garber AJ, Kim DK. Fenofibrate lowers abdominal and skeletal adiposity and improves insulin sensitivity in OLETF rats. Biochem Biophys Res Commun. 2002 Aug 16;296(2):293-9. doi: 10.1016/s0006-291x(02)00822-7. PMID 12163016
- [Background] Idzior-Walus B, Sieradzki J, Rostworowski W, Zdzienicka A, Kawalec E, Wojcik J, Zarnecki A, Blane G. Effects of comicronised fenofibrate on lipid and insulin sensitivity in patients with polymetabolic syndrome X. Eur J Clin Invest. 2000 Oct;30(10):871-8. doi: 10.1046/j.1365-2362.2000.00734.x. PMID 11029601
- [Background] Yong QW, Thavintharan S, Cheng A, Chew LS. The effect of fenofibrate on insulin sensitivity and plasma lipid profile in non-diabetic males with low high density lipoprotein/dyslipidaemic syndrome. Ann Acad Med Singap. 1999 Nov;28(6):778-82. PMID 10672386